CLINICAL TRIAL: NCT01015521
Title: A Two-Arm Open Label Phase II Study of AFP464 (Aminoflavone Prodrug) in Previously-treated ER-positive or Triple-negative Breast Cancer Patients
Brief Title: Efficacy Study of Aminoflavone Prodrug to Treat Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated as planned
Sponsor: Tigris Pharmaceuticals (Industry)
Responsible Party: Binh Nguyen, MD PhD, Chief Medical Officer
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-AFP-002
Record Dates: First submitted 2009-11-16; First posted 2009-11-18 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Breast Neoplasm
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aminoflavone Prodrug (Experimental): Aminoflavone to treat ER positive breast cancer patients
  Interventions: Drug: Aminoflavone Prodrug
- Aminoflavone Prodrug with pretreatment (Experimental): Aminoflavone Prodrug to treat Triple Negative Breast Cancer
  Interventions: Drug: Aminoflavone Prodrug

INTERVENTIONS:
Drug: Aminoflavone Prodrug — Aminoflavone Prodrug administered D1, D8 of 21-day cycle
  Other Names: AFP464

SUMMARY:
This is a phase II study to assess the efficacy of Aminoflavone prodrug in triple negative and ER+ breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* ER+ or TN Breast Cancer
* Progression on an aromatase inhibitor if ER+
* Prior treatment with taxane if TN
* 18 years or older
* Adequate organ function
* Measurable lesion

Exclusion Criteria:

* symptomatic pulmonary disease
* brain metastases
* pregnant females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Benefit Response | 6 months

SECONDARY OUTCOMES:
Progression Free Survival | 6 monhts

REFERENCES:
- [Derived] Saito R, Miki Y, Hata S, Ishida T, Suzuki T, Ohuchi N, Sasano H. Aryl hydrocarbon receptor induced intratumoral aromatase in breast cancer. Breast Cancer Res Treat. 2017 Feb;161(3):399-407. doi: 10.1007/s10549-016-4063-x. Epub 2016 Nov 30. PMID 27900579